CLINICAL TRIAL: NCT00019214
Title: Phase I/II Study in Patients With Metastatic Melanoma of Immunization With Dendritic Cells Presenting Epitopes Derived From The Melanoma Associated Antigens MART-1 and gp 100
Brief Title: Vaccine Therapy With or Without Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065234; NCI-97-C-0046; NCI-97-C-0019; NCI-T96-0046N; NCT00001558 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2005-01

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; aldesleukin

INTERVENTIONS:
Biological: MART-1 antigen
Biological: aldesleukin
Biological: gp100 antigen

SUMMARY:
RATIONALE: Vaccines made from white blood cells treated with antigens may make the body build an immune response to kill melanoma cells. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Combining vaccine therapy with interleukin-2 may kill more melanoma cells.

PURPOSE: This phase I/II trial is studying the side effects and how well giving vaccine therapy and interleukin-2 works compared to vaccine therapy alone in treating patients with metastatic melanoma that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the toxicity, immunologic reactivity, and possible therapeutic efficacy of immunization with dendritic cells presenting the MART-1 and gp100 melanoma antigens with or without interleukin-2 in patients with metastatic melanoma.

OUTLINE: This is a dose-escalation study of dendritic cells pulsed with MART-1 and gp100 antigens.

Patients receive vaccinations with dendritic cells pulsed with MART-1 and gp100 antigens, either intralymphatically every 4 weeks for 2 doses, or IV every 3 weeks for 4 doses. Some patients also receive interleukin-2 subcutaneously or IV, over 3-5 days, beginning 24 hours after immunization.

Cohorts of 2-9 patients receive escalating doses of pulsed dendritic cells IV until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Subsequent cohorts receive cells with or without interleukin-2. One cohort may expand to 15 patients to determine the accuracy of immunologic response to the vaccine.

One cohort of 11 patients receives cells intralymphatically without interleukin-2 every 3-4 weeks for 2 courses. Patients with stable disease or who achieve minor, mixed, or partial response may be retreated.

Patients with stable or responding disease undergo a second course of vaccination. Patients who completed treatment with vaccine alone and have stable disease, progressive disease, disease progression after a response, or a partial response with no further improvement may receive 2 additional courses.

PROJECTED ACCRUAL: A total of 10-42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma that has failed standard effective therapy
* Measurable or evaluable disease
* HLA-A2 positive

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8.0 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST/ALT less than 4 times upper limit of normal
* Negative hepatitis B surface antigen
* No coagulation disorder

Renal:

* Creatinine no greater than 1.6 mg/dL OR
* Creatinine clearance greater than 75 mL/min

Cardiovascular:

* No major cardiovascular disease

Pulmonary:

* No major respiratory disease

Other:

* No major immunological disease
* No penicillin allergy
* HIV negative
* No active systemic infection
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* At least 4 weeks since prior steroid therapy and recovered

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 4 weeks since any other prior therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-04; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Yang, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States